CLINICAL TRIAL: NCT07123636
Title: A Clinical Study to Assess the Effect of Hair Care Products on Grey Hair and Overall Hair Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Two Lines LLC (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20385
Record Dates: First submitted 2025-04-22; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hair Aging; Hair Graying
Keywords: Hair Health; Hair Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hair Care Products (Experimental): All participants will receive the four products and use them as directed over 24 weeks.
  Interventions: Dietary Supplement: Hair Care Products

INTERVENTIONS:
Dietary Supplement: Hair Care Products — Daily oral intake of 2 tablets (Not Today, Grey). Twice-daily application of 3-4 pumps of "To The Root" serum. Wash and Smooth used according to hair type (daily or every other day).

SUMMARY:
This is a 24-week virtual, single-arm study designed to evaluate the effectiveness of a hair care system-comprising the "Not Today, Grey" supplement, "To the Root" scalp serum, "Wash" shampoo, and "Smooth" conditioner-on grey hair reduction and overall hair health. Assessments include clinical grading of photographic evidence by dermatologists and participant-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (35% male and 65% female)
* Aged 25-55
* Must experience 5-25% of hair being grey as confirmed by a dermatologist grading of the baseline photo (see Figure 1 below)
* Any hair color that the investigator can clearly distinguish grey hairs from the natural hair color.
* Individuals who have not dyed or highlighted their hair for at least 6 months prior to screening/baseline and who agree to refrain from dyeing the hair until after the final study visit.
* Willing to maintain the same hairstyle and length.
* Willing to refrain from using any topical hair products (other than Wash, Smooth, and To The Root) or treatments on the hair that could affect hair properties (e.g., heat treatments other than blowdrying, medicated shampoo) for the duration of the study.
* Willing to refrain from taking any vitamins, minerals, or herbal supplements with claims related to hair growth or benefits during the study and to not start taking any new vitamins, minerals, or supplements of any kind during the study.
* Willing to comply with the protocol, take all required photos, and immediately report any changes in health status or medications, adverse events, symptoms, or reactions.
* Willing and able to provide written informed consent, including an agreement to privacy language compliant with country and/or local requirements, after the scope and nature of the investigation have been explained and before the initiation of any study-related procedures.
* Must have a recent smartphone (iPhone 11 pro or greater/android equivalent).

Exclusion Criteria:

* Anyone with pre-existing conditions that would prevent participants from adhering to the protocol, including oncological, immunological, psychiatric disorders, uncontrolled diseases, or multiple controlled diseases.
* Anyone pregnant, trying to conceive, or breastfeeding.
* Anyone unwilling to follow the protocol.
* Anyone currently participating in another research study.
* Anyone with any known severe allergic reactions or with any allergies of any severity to any of the test product's ingredients (e.g., sesame).
* Anyone with a medical history of any condition that results in grey hair (for example, nutritional deficiencies, such as B12, iron, and copper deficiency, severe protein malnutrition, cystic fibrosis, celiac disease, hyperthyroidism/hypothyroidism, vitiligo, alopecia areata, and genetic diseases such as Werner syndrome, Louis-Bar syndrome, Waardenburg syndrome, or Griscelli syndrome).
* Having a medical history of any condition that results in hair darkening (e.g., Addison's disease, neurodermatitis, porphyria cutanea tarda, and inflammatory scalp conditions).
* Anyone currently receiving iron injections.
* Anyone who is currently a smoker or has smoked regularly in the last six months.
* Anyone who has a history of substance abuse (i.e., within six months prior to screening).
* Anyone who has started long-term medication within the last two months.
* Anyone who is having any planned surgeries or invasive procedures during the study period (24 weeks) or has undergone an invasive procedure three weeks prior to the study start.
* Anyone who has used an investigational drug or device within the 30 days prior to screening.
* Anyone who is currently undergoing hormone therapy (e.g., HRT, or testosterone) and anyone who in the last three months has undergone hormone therapy.

Ages: 25 Months to 55 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Grey Hair Assessed by Dermatologists | Baseline, Week 12, Week 24
  Assessment of photographic evidence (baseline, week 12, and week 24) to evaluate reduction in grey hair. Two trained dermatologists will review photos in a blinded order and answer yes/no questions on greying reduction and repigmentation.

SECONDARY OUTCOMES:
Participant Self-Reported Changes in Hair Health | Weeks 6, 12, 18, and 24
  Participants will complete questionnaires assessing their perception of grey hair amount, hair softness, shine, texture, strength, thickness, and overall hair quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No